CLINICAL TRIAL: NCT06890442
Title: Associated Radiological Variations in the Skull Bones in Patients with Cong: Unilateral Choanal Atresia
Brief Title: Skull Bon Variations in Patient with Congenital Unilatral Choanal Atresia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Sayed Mohamed Moaz, Principal investigator, Assiut University
Other Study IDs: Skull bon in CUCA patient
Record Dates: First submitted 2025-03-06; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CT — Thickened Medial Pterygoid Plates In bony atresia, excessive thickening of the medial pterygoid plates is common. Narrowing or Fusion of the Posterior Choanae Complete bony or membranous obstruction at the choanal opening. Abnormal Sphenoid Bone Development Hypoplasia or deformity in the sphenoid sinus, affecting adjacent structures. Vomer Deviation or Hypertrophy The vomer bone is often displaced or abnormally thickened, contributing to obstruction.
  Abnormal Development of the Hard Palate

SUMMARY:
Identify skull bone Associated Anomalies in patients with cngenital unilatral choanal atresia

DETAILED DESCRIPTION:
Choanal atresia is a rare congenital disorder caused by a failure to develop the posterior nasal cavity (choana), resulting in a missing opening between the nasopharynx and the nasal cavities.It is the most common congenital anatomical abnormality of the nasal cavities with incidence ratio approximately 1/5000-7000 live births

Generally, choanal atresia may affect one or both Choanae, although most studies show that the unilateral form is more common than the bilateral one,and the incidence is higher in females than in males Children with unilateral choanal atresia are subject to unilateral breathing usually have late unilateral nasal obstruction, persistent ipsilateral rhinorrhea, and recurrent rhinosiusitis Previous studies have shown that the ratio of bone to membranous atresia is 9:1; although a detailed review of CT findings with histopathological studies showed that mixed-wall atresia is the most common and is present in 71% of cases, while in 29% of cases we found a pure bone wall Computer tomography (CT) is presently the golden standard in diagnostics of nasal cavity diseases; thus, it can be applied successfully as a tool for assessing anatomical structures

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Congenital Unilateral Choanal Atresia

Exclusion Criteria:

Patients with severe craniofacial syndromes

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients diagnosed with congenital unilateral choanal atresia (CUCA). The inclusion and exclusion criteria will ensure a well-defined and homogenous group for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Radiological Variations in Skull Bones in Patients with Congenital Unilateral Choanal Atresia: A Cross-Sectional Study" | 10_12 month
  Degree and Type of Skull Bone Anomalies Presence and extent of bony abnormalities in the skull base (e.g., sphenoid bone asymmetry, pterygoid plate thickening) Degree of nasal cavity narrowing and choanal obstruction Associated maxillofacial bone abnormalities (e.g., septal deviation, maxillary sinus hypoplasia)
  2. Measurement of Specific Skull Bone Changes
  Thickness of the atretic plate (bony vs. membranous) Asymmetry of pterygoid plates (measured in mm) Deviation angle of the nasal septum (in degrees) Orbital and maxillary asymmetry

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ragab Sayed, Lecturer, Principal Investigator

REFERENCES:
- [Background] Kwong KM. Current Updates on Choanal Atresia. Front Pediatr. 2015 Jun 9;3:52. doi: 10.3389/fped.2015.00052. eCollection 2015. PMID 26106591